CLINICAL TRIAL: NCT05745428
Title: Shear Stress Endothelial/Hemodynamics in Aortic Dissection and Endothelial Shear Stress-biological Profile HADES-BP
Brief Title: Shear Stress Endothelial/Hemodynamics in Aortic Dissection and Endothelial Shear Stress-biological Profile
Acronym: HADES-BP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Pedicino Daniela, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4626
Record Dates: First submitted 2023-02-15; First posted 2023-02-27 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Aortic Dissection
Keywords: hypertension; vasospasm
MeSH Terms: conditions — Aortic Dissection; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — circulating biomarker analysis, aortic endothelial cell culture, peripheral whole blood collection and isolation of mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First group with aortic dissection: 19 patients admitted to our Department of Cardiovascular Sciences with a radiological diagnosis of AD within 14 days of the onset of symptoms
  Interventions: Other: molecular and cellular analyses
- Control Group: 19 healthy outpatient or inpatient controls at our Department with another diagnosis and no evidence of AD, matched for demographic and clinical characteristics.
  Interventions: Other: molecular and cellular analyses

INTERVENTIONS:
Other: molecular and cellular analyses — sample blood
  Other Names: Peripheral whole blood collection and isolation of mononuclear cells

SUMMARY:
Aortic dissection (AD) is a clinical condition belonging to the broader spectrum of Acute Aortic Syndromes, with high morbidity and mortality and characterised by the sudden formation of a breach within the tonaca intima of the aortic wall, from which the so-called false lumen originates.The most common risk factor for AD is hypertension, present in more than 70% of.

Imaging, biomarkers and genetic predisposition are critical in confirming a suspected diagnosis and in determining the appropriate intervention for each patient. Specific features influencing management decisions are the presence of rupture, extent of dissection, origin of true or false lumen vessels and signs of organ ischaemia.

DETAILED DESCRIPTION:
The aim of this study is to investigate the diagnostic value of circulating biomarkers and in aortic tissue in patients with AD and to assess the prognosis of patients with AD and its complications in relation to the aforementioned markers, integrating biological data with clinical and instrumental data relating to the patient's hospitalisation.

The study involves a comparison between two arms, one experimental and the other control (healthy outpatients). A longitudinal evaluation will be carried out on the experimental arm with a follow-up visit (FUp) at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* partecipants admitted to our Department of Cardiovascular Sciences with a radiological diagnosis of AD within 14 days of the onset of symptoms;
* healthy outpatient or inpatient controls at our Department with another diagnosis and no evidence of AD, matched for demographic and clinical characteristics

Exclusion Criteria:

* evidence of inflammatory diseases, infectious diseases, neoplasms, immunological or haematological disorders;
* treatment with anti-inflammatory drugs with the exception of low-dose aspirin (75-160 mg);
* age > 85 years;
* advanced chronic kidney disease with glomerular filtration rate (eGFR) estimated by MDRD equation <30 ml/min./1.73 m2; 5) pregnancy;
* dissection with traumatic aetiology;
* failure to sign informed consent;

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants in this study present aortic dissection in its acute form (< 14 days) leading to short-term complications such as aortic rupture and visceral malperfusion, while the subacute (15-90 days) and chronic (> 90 days) forms lead to a process of aortic remodelling characterised by fibrinolysis and extracellular matrix (ECM) proteolysis, the latter being potential causes, in the long term, of gradual aortic dilatation with aneurysmal degeneration.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2024-04-16 (Estimated)

PRIMARY OUTCOMES:
Evaluation of gene expression | 1 year
  Evaluation of gene expression (by RT-qPCR),the analysis of circulating biomarkers smMYO11 (Human Myosin Heavy Chain 11, SmoothMuscle (MYH11) ELISA Kit, My Biosource), Calponin (Human Calponin-1 ELISA Kit, My Biosource) and MMP-9 (Human MMP-9 Quantikine ELISA Kit, R&D System ) will be performed by enzyme immunoassay on suitably preserved serum from AD and CTRL partecipants, in accordance with the manufacturer's instructions.
Evaluation of transcriptomics | 1 year
  This study will be perfomed by single-cell analysis with enzyme immunoassay thanks to the peripheral blood sample that was taken from the participant at the time of enrollment
Evaluation of protein | 1 year
  This evaluation immunoenzymatic analyses, it's important to analyze altered biomarkers following fluid dynamic alterations applied by controlled mechanical stress to a model of primary cultures of aortic endothelial cells (HAOEC) and peripheral mononuclear cells (PBMC) isolated from enrolled subjects.

SECONDARY OUTCOMES:
Assessment of correlation between circulating biomarkers | 1 year
  Assessment of correlation between circulating biomarkers, clinical data (signs of haemodynamic stability such as blood pressure (BP), heart rate (HR), oxygen saturation (SpO2), signs of organ malperfusion such as neurological signs distal pulses, oligo-anuria or signs of outward rupture such as cardiac tamponade, acute aortic valvular insufficiency, haemothorax, haemoperitoneum), and imaging data (diameter of the ascending aorta ≥5 5cm, intimal breach size >10mm, diameter of the false lumen >22mm, partial thrombosis of the false lumen, intimal flap concave towards the false lumen, periaortic haematoma, single entry port or localisation of this in the small curvature of the aortic arch)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy